CLINICAL TRIAL: NCT04472260
Title: Early Verticalization of the Patient With Acute Respiratory Distress Syndrome: Assessment of Feasibility and Safety.
Acronym: STAND_ARDS1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CHRO-2018-12
Record Dates: First submitted 2020-06-25; First posted 2020-07-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome; Prone Position
Keywords: Acute respiratory distress syndrome; Verticalization; Intensive Care Unit; Prone position
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: In order to compare the effect of prone position (PP) and verticalization (V) on the PaO2/FiO2 ratio (secondary objective of the study), a randomized cross-over experimental design was chosen.
  Patients will be randomly assigned to one of the following 4 sequences. They will each include 4 treatment periods:
  Sequence 1: PP->PP->V->V, Sequence 2: PP->V->V->PP, Sequence 3: V->PP->PP->V Sequence 4: V->V->PP->PP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1: PP->PP->V->V (Other): The randomly selected study sequence (Arm1, Arm2, Arm3 or Arm4) will begin after the supine roll-over at the end of the first PP session (out-of-study sequence). This allows all patients to initially have the positioning technique that has been proven beneficial in ARDS.
  The chronology of the treatment periods in each of the 4 arms allocated by randomization will be as follows: Each PP must be started within 4 to 8 hours after the end of the previous PP or after the end of the verticalization that just preceded it. Each verticalization must be performed within 4 to 8 hours after the end of the previous PP or the previous verticalization. Each PP period will last between 12 and 20 hours.
  Interventions: Procedure: Verticalization and Prone position
- Sequence 2: PP->V->V->PP (Other): The randomly selected study sequence (Arm1, Arm2, Arm3 or Arm4) will begin after the supine roll-over at the end of the first PP session (out-of-study sequence). This allows all patients to initially have the positioning technique that has been proven beneficial in ARDS.
  The chronology of the treatment periods in each of the 4 arms allocated by randomization will be as follows: Each PP must be started within 4 to 8 hours after the end of the previous PP or after the end of the verticalization that just preceded it. Each verticalization must be performed within 4 to 8 hours after the end of the previous PP or the previous verticalization. Each PP period will last between 12 and 20 hours.
  Interventions: Procedure: Verticalization and Prone position
- Sequence 3: V->PP->PP->V (Other): The randomly selected study sequence (Arm1, Arm2, Arm3 or Arm4) will begin after the supine roll-over at the end of the first PP session (out-of-study sequence). This allows all patients to initially have the positioning technique that has been proven beneficial in ARDS.
  The chronology of the treatment periods in each of the 4 arms allocated by randomization will be as follows: Each PP must be started within 4 to 8 hours after the end of the previous PP or after the end of the verticalization that just preceded it. Each verticalization must be performed within 4 to 8 hours after the end of the previous PP or the previous verticalization. Each PP period will last between 12 and 20 hours.
  Interventions: Procedure: Verticalization and Prone position
- Saquence 4: V->V->PP->PP (Other): The randomly selected study sequence (Arm1, Arm2, Arm3 or Arm4) will begin after the supine roll-over at the end of the first PP session (out-of-study sequence). This allows all patients to initially have the positioning technique that has been proven beneficial in ARDS.
  The chronology of the treatment periods in each of the 4 arms allocated by randomization will be as follows: Each PP must be started within 4 to 8 hours after the end of the previous PP or after the end of the verticalization that just preceded it. Each verticalization must be performed within 4 to 8 hours after the end of the previous PP or the previous verticalization. Each PP period will last between 12 and 20 hours.
  Interventions: Procedure: Verticalization and Prone position

INTERVENTIONS:
Procedure: Verticalization and Prone position — The randomly selected study sequence (Arm1, Arm2, Arm3 or Arm4) will begin after the supine roll-over at the end of the first PP session (out-of-study sequence). This allows all patients to initially have the positioning technique that has been proven beneficial in ARDS.
  The chronology of the treatment periods in each of the 4 arms allocated by randomization will be as follows: Each PP must be started within 4 to 8 hours after the end of the previous PP or after the end of the verticalization that just preceded it. Each verticalization must be performed within 4 to 8 hours after the end of the previous PP or the previous verticalization. Each PP period will last between 12 and 20 hours.

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is defined according to the Berlin definition (1) as diffuse lung damage occurring in patients with a predisposing risk factor.

Positioning in the prone position (PP) has been shown to decrease mortality in patients with moderate to severe ARDS.

However, this technique is not without deleterious effects such as ventilator-associated pneumonia, endotracheal tube obstruction, development of pressure ulcers, and increased workload for the caregivers.

There are other positioning techniques such as the "upright" position, which simulates a relative verticality, which allows to increase the effects of the prone position and even in some patients to improve oxygenation without the PP in the acute phase of ARDS.

However, given the revolution caused by the use of PP in ARDS patients, verticalization have not been studied in more details.

Today, there is a bed on the market that allows patients to be truly upright without having to transfer them to a tilt table.

The investigators believe that raising ARDS patients in the acute phase is safe and feasible in routine practice. In this research protocol comparing PP and verticalization in a crossover trial design in acute ARDS patients, the investigators want to show that this technique can be safe and feasible, with the same effects on oxygenation as PP.

DETAILED DESCRIPTION:
Cross-over study, according to 4 preset sequences of 4 periods and randomly assigned. All patients will thus have the classic positioning technique (PP), as well as the technique under study (verticalization). For simplicity, the investigators will use the term "verticalization" even if the final positioning that is targeted is only a "pseudo-verticalization" to a 55° angle. The cross-over scheme with 4 sequences of 4 periods allows to get rid of the first order carry-over effect.

Progressive verticalization protocol in 7 steps from the strict supine position to a 55° inclination of the raising bed, according to the clinical responses of the patient with ARDS, as follows:

- Verticalization in the bed

The verticalization maneuver will take place in 7 steps of 15 minutes maximum each:

S1. The first one corresponds to the flat position (strict dorsal decubitus) S2. The second is the positioning of the patient at 25° of inclination. S3. The third is the 45° positioning S4. The fourth at 55°, which corresponds to the greatest inclination imposed to the patient.

S5. The fifth corresponds to the 45° return S6. The sixth is the return to 25° S7. Finally, the investigators reposition the patient flat back.

Examinations:

* Arterial Gazometry At the beginning, at the end and one hour after each positioning technique.
* Chest ultrasound
* Others All adverse events will be recorded in a clear and detailed manner.

ELIGIBILITY:
Inclusion Criteria:

* Major patient > 18 years of age
* ARDS patients with PaO2/FiO2 ratio < 150 at any time within 24 hours prior to the screening visit
* Hemodynamically stable patient with mean arterial pressure (MAP) > 65 mmHg maintained without vasopressor or with norepinephrine at a dosage of less than 0.5 µg/kg/min.
* Patient having already undergone at least 1 but less than 5 PP sessions
* Patient under continuous intravenous sedation (IVSE) or not responding to simple order.
* Written consent of support person or family.

Exclusion Criteria:

* Pregnant women (positive pregnancy test during screening)
* Breastfeeding women
* Protected Majors
* Body weight greater than 198 kg (bed load limit)
* Patient with one or two lower limbs amputated at the trans tibial or upper level
* Contraindication to standing (orthopedic fracture, neurological instability with the presence of an intracranial pressure sensor or an external ventricular shunt....)
* Deep venous thrombosis of the lower limbs with curative anticoagulation for less than 48 hours
* Hemodynamic instability (MAP < 65 mm Hg) despite the use of norepinephrine at a dosage equal or greater than 0.5 µg/kg/min.
* Person under guardianship or trusteeship
* Non-beneficiary patient of a health insurance plan
* Moribund patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who were able to reach 55° of verticalization without serious adverse events (with a complete listing of all adverse events). | Month 1
  To demonstrate the feasibility and safety in routine practice of the verticalization technique for patients with moderate to severe ARDS in the acute phase.

SECONDARY OUTCOMES:
PaO2/FiO2 ratio at one hour from the end of the maneuver | Hour 76
  To show that verticalization of ARDS patients has the same effects on oxygenation (PaO2/FiO2 ratio) as PP.
  In this crossover trial, each sequence of four treatment periods, beginning at time of randomization, will last a maximum of 75,5 hours for each patient. The last assessment will occur at a maximum of 76,5 hours from randomisation.
Quasi-static compliance in (ml/cmH2O) before, at the end and one hour after each positioning technique | Hour 76
  To evaluate the impact of the positioning maneuver on quasi-static thoracopulmonary compliance.
  In this crossover trial, each sequence of four treatment periods, beginning at time of randomization, will last a maximum of 75,5 hours for each patient. The last assessment will occur at a maximum of 76,5 hours from randomisation.
Lung Reaeration Score at 1 hour from the end of the maneuver | Hour 76
  To compare the re-ventilation of the pulmonary territories at one hour of the session (PP or verticalization) evaluated by thoracic ultrasound.
  In this crossover trial, each sequence of four treatment periods, beginning at time of randomization, will last a maximum of 75,5 hours for each patient. The last assessment will occur at a maximum of 76,5 hours from randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Mai-ANh NAY, Dr, Principal Investigator — CHR Orléans
Locations (1):
- CHR d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Umbrello M, Formenti P, Bolgiaghi L, Chiumello D. Current Concepts of ARDS: A Narrative Review. Int J Mol Sci. 2016 Dec 29;18(1):64. doi: 10.3390/ijms18010064. PMID 28036088